CLINICAL TRIAL: NCT01264627
Title: Project Inspire: A New Translational Tool for Studying the Role of Breathing in Meditation
Brief Title: A New Translational Tool for Studying the Role of Breathing in Meditation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01AT005820 (NIH); 1R01AT005820 (NIH)
Record Dates: First submitted 2010-12-15; First posted 2010-12-22 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure; Breathing; PetCO2; Stress
MeSH Terms: conditions — Hypertension; Respiratory Aspiration | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindful Breathing (MB) (Experimental): The MB intervention is based off of the Mindfulness Based Stress Reduction Program developed by Jon Kabat-Zinn. Participants will be organized into cohorts of eight, and attend eight weekly MB sessions. Mindful breathing consists of closely "following the breath," throughout inhalation and exhalation, sustaining moment-to-moment awareness on the breathing process, and passively observing thoughts, affective states, perceptions and events, from a non-evaluative, non-judgmental perspective. No other intervention is included. No FDA drug or device is involved.
  Interventions: Behavioral: Mindful Breathing (MB) Intervention
- Usual Care (UC) (Other): Usual Care consists of the standard care made available to participants through their primary physician. No intervention is included. No FDA drug or device is involved.
  Interventions: Behavioral: Usual Care (UC) Control Condition

INTERVENTIONS:
Behavioral: Mindful Breathing (MB) Intervention — The Mindful Breathing (MB)intervention is based on MBSR developed by Jon Kabat-Zinn. Participants will attend 8 individual weekly MB sessions. MB consists of closely "following the breath," throughout inhalation and exhalation, sustaining moment-to-moment awareness on the breathing process, and passively observing thoughts, affective states, from a non-evaluative or judgmental perspective. As attention wanders to concerns or thoughts, participants will be instructed to acknowledge and accept these without evaluation and return the focus of attention back to breathing. Participants in MB will have their breathing rate and PetCO2 monitored during the 8 training sessions with a breathing monitor.
  Arms: Mindful Breathing (MB)
Behavioral: Usual Care (UC) Control Condition — This control intervention is designed to account for the effects of nonspecific factors such as enrollment in a study to enhance health with the associated expectancy effects, staff attention, and measurement procedures including the monitoring of PetCO2 and (Blood Pressure) BP, and completion of questionnaires. Participants who are randomly assigned to the Usual Care condition will receive care as usual for the management of their prehypertensive condition. UC participants will receive their usual care and have access to all Kaiser Permanente (KP) health education resources, such as KP's interactive healthcare guide, and online "Healthy Lifestyle Programs". We will assess the extent to which participants in both MB and UC used these resources.
  Arms: Usual Care (UC)

SUMMARY:
A recent National Health Interview Survey reported that breathing exercises were the second most common complementary and alternative medicine practice in the United States, following only the use of "natural products." With such widespread interest in breathing exercises, alone or as a component of practices such as meditation, a need exists for research that examines not only its efficacy, but also investigates potential mechanisms of action. Indeed, a recent National Center for Complementary and Alternative Medicine (NCCAM) Meditation Workshop recommended research to clarify biological pathways by which meditation practices, including breathing exercises, can impact health. To explore mechanisms underlying the health effects of breathing exercises, new translational tools are needed that can measure breathing patterns in both the clinic and natural environment. The primary objective of the present proposal is the application of a new technology to the investigation of pathways by which breathing exercises can affect health. For this project, the health-related outcome measure to be studied is a major cardiovascular risk factor, blood pressure.

ELIGIBILITY:
Inclusion Criteria

* Mean 24-hr SBP: 130-139 mmHg
* Female
* > 50 years of age
* Post menopausal, defined as greater than or equal to one year without a menstrual cycle.
* Body Mass Index (BMI): 19-31
* English speaking (Patients not able to read and speak English will be excluded as the behavioral group interventions are conducted in English)
* Has a personal physician

Exclusion Criteria (Individuals will be filtered in the KP OSCA database according to the following ICD-9 codes):

Respiration:

* 491.X chronic Bronchitis incl COPD
* 492.X emphysema
* 493.X asthma
* 494-496; 500-519: all kinds of chronic pulmonary conditions

Cardiovascular:

* 404.9 chronic ischemic heart disease
* 425.X cardiomyopathies
* 428.X heart failure
* 430-438 cerebrovascular diseases

Kidney:

* 582-583 chronic glomerulonephritis
* 584-588 renal failure

Liver:

- 571.X chronic liver disease and cirrhosis Smoker: 305.1

Psychiatric:

* 290-299 dementia/schizophrenia/ psychoses…
* 303, 304 alcohol or drug dependence
* 317-319 mental retardation

Medications:

* All blood pressure medications
* All tranquilizers, benzodiazepins if prescribed regularly, e.g. every month
* All narcotics if prescribed regularly, e.g. every month

Other:

- Plan to relocate residence outside recruitment area during the intervention or follow- period

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Up to Week 25
  Measured using Ambulatory, 24-Hr BP monitor

SECONDARY OUTCOMES:
Clinic (resting) blood pressure | Up to Week 25

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A Chesney, PhD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnes PM, Bloom B, Nahin RL. Complementary and alternative medicine use among adults and children: United States, 2007. Natl Health Stat Report. 2008 Dec 10;(12):1-23. PMID 19361005